CLINICAL TRIAL: NCT00621816
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Determine the Pharmacodynamics of Sodium Nitroprusside During Prolonged Infusion in Pediatric Subjects
Brief Title: Sodium Nitroprusside for Blood Pressure Reduction in the ICU (SNP2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: N01-HD-4-3386; NICHD-2003-09-DR
Record Dates: First submitted 2008-02-20; First posted 2008-02-22 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: nitroprusside; intensive care unit; hypertension; blood pressure reduction
MeSH Terms: conditions — Hypertension | interventions — Nitroprusside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Blinded nitroprusside infusion
  Interventions: Drug: nitroprusside
- 2 (Placebo Comparator): Blinded placebo infusion
  Interventions: Drug: placebo infusion

INTERVENTIONS:
Drug: nitroprusside — nitroprusside continuous infusion, dose to be titrated to clinical effect
  Other Names: Nipride
  Arms: 1
Drug: placebo infusion — blinded placebo infusion, to be infused at same rate as open-label nitroprusside infusion
  Arms: 2

SUMMARY:
Nitroprusside is used commonly in the Intensive Care Unit for long periods of time in order to reduce blood pressure. It is not known if the body compensates over time to the blood pressure lowering, and if when the nitroprusside is stopped the blood pressure goes up at a faster rate and is higher than it was at the start of the treatment. This study will answer these questions.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, randomized, double-blind placebo-controlled, parallel group study to determine the persistence of the effect of SNP on blood pressure and to assess the potential for rebound hypertension associated with prolonged infusion in pediatric subjects.

The primary endpoint is the change in MAP during the Blinded Study Drug Administration Phase in the absence of other stimuli.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is less than 17 years of age.
2. An in-dwelling arterial line is clinically indicated.
3. Subject's parent or legal guardian is willing and able to give informed parental permission signing and dating an IRB-approved informed parental permission containing all of the elements of informed consent, and subject provides assent, signing an IRB-approved and -required informed assent, if applicable.
4. Subject is anticipated to require a minimum of 20 mm Hg (15 mm Hg for subjects < 2 years old) reduction in MAP for at least 12 hours using SNP [i.e., MAPB1 - MAPB2 ≥ 20 mm Hg (15 mm Hg for subjects < 2 years old)]

Exclusion criteria:

1. Subject weighs < 3.0 kg.
2. Subject has a known allergy to SNP.
3. Subject has a known mitochondrial cytopathy with a disorder of oxidative phosphorylation or of respiratory chain enzymes.
4. Subject has a contraindication to vasodilator therapy for control of blood pressure during surgery or in the intensive care unit.
5. Subject has raised intracranial pressure.
6. Subject is anticipated to need anti-hypertensive drugs other than Sodium Nitroprusside either IV (e.g. dexmedetomidine, esmolol, etc.) or epidural (e.g.local anesthetics, clonidine, etc.) within three terminal half-lives (3X T½ β) of the blinded study drug period. However, patients receiving stable doses of an anti-hypertensive drug(s) prior to the initiation of study drug may be enrolled.
7. Subject has any serious medical condition which, in the opinion of the investigator, is likely to interfere with study procedures.
8. Subject is moribund (death likely to occur within 48 hours).
9. Subject has a positive result for the urine or serum HCG test administered at screening.
10. Subject has participated in other clinical trials for investigational drugs within 30 days prior to enrollment
11. Subject has received or will have received Sodium Thiosulfate within 6 hours prior to the start of the open-label period.
12. Subject is either on, or anticipated to be on, ECMO.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in MAP during the Blinded Study Drug Administration Phase in the absence of other stimuli. | 8 months

SECONDARY OUTCOMES:
1. To compare the proportion of patients randomized to receive either sodium nitroprusside or placebo who experience offset during the 30-minute blinded study drug period. | 8 months
2. To compare the proportion of patients randomized to receive either sodium nitroprusside or placebo who experience rebound hypertension during blinded study drug period | 8 months
3. To compare the proportion of patients randomized to receive either sodium nitroprusside or placebo who experience a serious adverse event during the 30-minute blinded study drug period | 8 months
4. To compare the distribution of patients randomized to receive either sodium nitroprusside or placebo who experience a treatment-emergent and related adverse event, by maximum severity grade, during the 30-minute blinded study drug period. | 8 months
5. To compare the changes in vital signs (systolic blood pressure, diastolic blood pressure, MAP, and heart rate) between patients randomized to receive either sodium nitroprusside or placebo | 8 months
6. To compare the changes in individual laboratory parameters between patients randomized to receive either sodium nitroprusside or placebo. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott Schulman, MD, Principal Investigator — Duke University; Greg Hammer, MD, Principal Investigator — Stanford University
Locations (7):
- United States (7):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Stanford University School of Medicine, Stanford, California
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - University of Michigan - Mott Children's Hospital, Ann Arbor, Michigan
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - West Virginia University, Morgantown, West Virginia